CLINICAL TRIAL: NCT01977105
Title: Abbreviated Pilot Trial of a Peer-Based Social Media Intervention to Promote Healthy Growth During Infancy
Brief Title: Healthy Growth Abbreviated Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-009905
Record Dates: First submitted 2013-09-30; First posted 2013-11-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Childhood Obesity
Keywords: Infants; Mothers; Social media; Obesity prevention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot Intervention Group (Experimental): Mothers who are screened and determined to be eligible for this single-group pilot study will be enrolled along with their infants in the Grow Together peer group intervention.
  Interventions: Behavioral: Grow Together peer group

INTERVENTIONS:
Behavioral: Grow Together peer group — Participants in this intervention will:
  * Participate in Facebook group of 6-10 peers for about 8 weeks, led by a professional group mentor.
  * Complete an intervention video activity approximately weekly:
    * 1. View educational videos addressing topics related to healthy infant growth
    * 2. Create photos/videos modeling healthy behaviors and post them to the group
    * 3. Provide and receive feedback on posts
    * 4. Be encouraged to share information with key caregivers of their child
  * Attend group party soon after enrollment, to meet peers and group leader in person.
  * Receive text message reminders, 1) to schedule recommended primary care visits for their infant, and 2) to attend appointments scheduled in CHOP Care Network.
  * Have basic program information provided to pediatrician to enhance conversation during office visits.

SUMMARY:
This is a single-group feasibility pilot trial of a peer-based, social media intervention to prevent obesity in infants.

DETAILED DESCRIPTION:
This novel intervention, delivered to mothers primarily through private Facebook groups, will promote behavior change through peer and self-modeling photo/video activities.

In this study, we will implement an abbreviated 2-month version of the intervention with a single peer group of up to 10 mothers. We will assess the feasibility and acceptability of both the intervention and our intended outcome measures, in preparation for a randomized pilot trial of the full intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years and older
* Enrolled in Medicaid at the time of study enrollment
* Overweight or obese (BMI >= 25, calculated using self-reported pre-pregnancy height and weight)
* Subjects able to speak, read and write in English
* Attend their infant's (up to 1 month old) primary care visit at a CHOP Primary Care Network site
* Received prenatal care
* Own a smartphone with both a data and text plan
* Able to use their phone to obtain photographs and videos prior to enrollment

Exclusion Criteria:

* Cannot provide consent.
* Non-English speaking.
* Score 10 or greater on Patient Health Questionnaire (PHQ-9) measure for clinical depression
* Diagnosed with gestational diabetes during pregnancy with their newborn
* Had a multiple pregnancy.
* Premature delivery (before 37 weeks) of their newborn.
* Have a newborn who was hospitalized in the Neonatal Intensive Care Unit (NICU) for one week or longer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability Survey | Study end (approximately 2 months)
  Satisfaction with the overall intervention will be assessed for mothers using a standard survey. Subjects will be asked a series of open-ended and Likert-scaled questions.
Study population eligibility and interest | Study end (approximately 2 months)
  * Proportion of all mothers contacted who meet enrollment criteria
  * Proportion of mothers meeting enrollment criteria who enroll
  These proportions will be calculated using study recruitment records.
Participant engagement | Study end (approximately 2 months)
  * Proportion of enrolled mother-infant dyads that comply with intervention participation requirements
  * Proportion of enrolled mother-infant dyads that complete each weekly module activity
  * Proportion of enrolled mother-infant dyads that complete each study measure
  * Number and type of each participant's Facebook group interactions per week (posts, comments, "Likes")
  * Frequency, type, and content of each contact between moderator/study staff and each participant
  This study process data will be obtained from the Facebook group and study records at study end.
Week 1 Curriculum Module Acceptability Survey | 1 week (approximately)
  Subjects will assess the Week 1 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 2 Curriculum Module Acceptability Survey | 2 weeks (approximately)
  Subjects will assess the Week 2 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 3 Curriculum Module Acceptability Survey | 3 weeks (approximately)
  Subjects will assess the Week 3 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 4 Curriculum Module Acceptability Survey | 4 weeks (approximately)
  Subjects will assess the Week 4 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 5 Curriculum Module Acceptability Survey | 5 weeks (approximately)
  Subjects will assess the Week 5 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 6 Curriculum Module Acceptability Survey | 6 weeks (approximately)
  Subjects will assess the Week 6 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 7 Curriculum Module Acceptability Survey | 7 weeks (approximately)
  Subjects will assess the Week 7 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.
Week 8 Curriculum Module Acceptability Survey | 8 weeks (approximately)
  Subjects will assess the Week 8 curriculum activity module using a short (approximately 10-item) survey consisting of Likert-scaled and open-ended questions.

OTHER OUTCOMES:
Infant feeding beliefs | Study start (enrollment to approximately 1 week) and study end (approximately 8 weeks)
  Maternal beliefs regarding infant feeding will be measured using the Infant Feeding Style Questionnaire (IFSQ), which contains 10 items measuring beliefs, coded on a 5-point scale (disagree, slightly disagree, neutral, slightly agree, agree).
Infant feeding practices | Study start (enrollment to approximately 1 week) and study end (approximately 8 weeks)
  Maternal behaviors related to infant feeding will be measured using 10 items on the Infant Feeding Style Questionnaire (IFSQ). Behavior items are coded on a 5-point scale (never, seldom, half of the time, most of the time, always).
  Also, four items from the validated Infant Feeding Practices Questionnaire (IFPQ) will be used to assess maternal feeding practices related to obesity. The IFPQ contains 20 items, with a 5-point adapted Likert response scale ranging from 0 (Never) to 4 (Always).
Breastfeeding survey | Study start (enrollment to approximately 1 week) and study end (approximately 8 weeks)
  Breastfeeding intent, initiation, and duration will be assessed using a survey
Introduction of solid foods and sugar-sweetened beverages | Study end (approximately 8 weeks)
  Timing of initiation of solid foods and sugar sweetened beverages will be assessed using a survey.
Infant sleep behaviors | Study end (approximately 8 weeks)
  Infant sleeping and related maternal activities will be measured using the validated Brief Infant Sleep Questionnaire (BISQ). Subjects will complete the abbreviated 13-item BISQ (A-BISQ), as well as 2 additional questions from the expanded version (E-BISQ).
Parenting self-efficacy | Study end (approximately 8 weeks)
  The Karitane Parenting Confidence Scale (KPCS) is a 15-item validated scale that will be used to measure parenting self-efficacy. Questions assess the frequency of certain beliefs, skills and abilities related to successful parenting, measured using a 4-point response structure (No, hardly ever; No, not very often; Yes, some of the time; Yes, most of the time).
Positive parenting behaviors | Study end (approximately 8 weeks)
  Mothers will be assessed regarding specific parenting practices using the 10-item Infant/Toddler (IT) Home Observation for Measurement of the Environment (HOME) Inventory. Individual responses for each yes/no item are coded to 0 or 1.
Maternal self-care behaviors | Study end (approximately 8 weeks)
  Mothers will be asked 11 questions related to their self-care behaviors, including their own sleep habits, support-seeking behaviors, and taking time for themselves. These items are a combination of Likert-scaled items and simple measures of the frequency of behaviors.
Maternal social support | Study start (enrollment to approximately 1 week) and study end (approximately 8 weeks)
  Mothers' level of social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). This validated scale is made up of 12 items. Responses for this scale are coded from 1 to 7 (very strongly disagree, strongly disagree, mildly disagree, neutral, mildly agree, strongly agree, and very strongly agree).
Maternal stress | Study end (approximately 8 weeks)
  The Parental Stress Scale (PSS) is a validated, 18-item public domain scale measuring perceived parental stress using a 5-point Likert rating scale ('Strongly disagree' to 'strongly agree').
Infant weight and growth | Study start (enrollment visit) and study end (approximately 8 weeks)
  Infants' weight will be measured using using a calibrated digital scale and length will be measured using a standard infantometer. Measurements will be taken by a trained nurse or other trained staff member at the primary care recruitment sites, or by a member of the study staff trained in anthropometric measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gruver RS, Bishop-Gilyard CT, Lieberman A, Gerdes M, Virudachalam S, Suh AW, Kalra GK, Magge SN, Shults J, Schreiner MS, Power TJ, Berkowitz RI, Fiks AG. A Social Media Peer Group Intervention for Mothers to Prevent Obesity and Promote Healthy Growth from Infancy: Development and Pilot Trial. JMIR Res Protoc. 2016 Aug 2;5(3):e159. doi: 10.2196/resprot.5276. PMID 27485934